CLINICAL TRIAL: NCT05138250
Title: A Pilot Study of the Use of 129Xe and 1H MRI to Measure the Modulation of Eosinophil-Related Inflammation by Mepolizumab In COPD
Acronym: SUMMER
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH21067
Record Dates: First submitted 2021-11-05; First posted 2021-11-30 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: COPD
Keywords: MRI, eosinophil, exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (all participants, not randomised) (Experimental): All participants will be treated with mepolizumab, a 100mg dose every 4 weeks for 1 year (13 doses)
  Interventions: Drug: Mepolizumab 100 MG

INTERVENTIONS:
Drug: Mepolizumab 100 MG — participants will receive 100mg of mepolizumab every 4 weeks for 52 weeks

SUMMARY:
The investigators aim to recruit 32 people with COPD who have frequent exacerbations and high eosinophil counts which indicates "asthmatic type" inflammation and treat them for a year with mepolizumab. This is a licenced medication for asthma. Mepolizumab is a monoclonal antibody that acts through interleukin-5 (IL-5) antagonism to reduce blood eosinophil levels and is effective at reducing exacerbations in asthmatics. To determine whether mepolizumab may be an effective treatment in people with COPD and "asthmatic type" inflammation participants will have MRI scans before the treatment, after 12 weeks and after a year to see how the drug affects inflammation. The investigators will also compare our measurements with the number of exacerbations people get (measured by diaries), with measures of their quality of life (using a questionnaire), and with ordinary laboratory breathing tests. The investigators are especially interested to know if the reduction in inflammation early on after 12 weeks is associated with fewer exacerbations and better quality of life over the year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD as determined by a post bronchodilator FEV1/FVC <70% and an FEV1 of between 20 and 80% at screening visit
* Treatment with inhaled triple therapy (licensed combination of long acting beta 2 agonist, long acting anti-muscarinic and corticosteroid) at constant dose for at least 12 weeks before screening visit. Treatment with roflumilast, theophyillines and macrolides will be permitted so long as they were introduced at stable dose > 12 weeks prior to screening visit. (If maintenance drug dosing has not been with stable dosages for 12 weeks the screening visit may be rescheduled until this is achieved: see sections 7.3 and 7.10)
* At least 2 acute exacerbations of COPD (AECOPD) requiring treatment with oral steroids and/or antibiotics in the last 12 months, or 1 acute AECOPD requiring hospital admission in the last 12 months.
* At least one eosinophil count of >0.3 cells·μL-1 in the 12 months prior to screening
* Age over 18 years

Exclusion Criteria:

* Contraindication to MRI scanning, including Gadovist (ie hypersensitivity or poor renal function; see below); this includes claustrophobia and musculoskeletal difficulties, this information is collected on the UoS MRI unit screening form.
* Inability to give informed consent or comply with study procedures
* Hypersensitivity to mepolizumab or its excipients
* Untreated helminthic infection
* Exacerbation of COPD requiring treatment with oral steroids and/or antibiotics within 4 weeks of screening. A repeat screening visit may be scheduled in order to achieve this criterion. The participant will be required to successfully complete all screening procedures at the rescheduled visit, including that for exacerbation-free stability.
* SpO2 <90% on room air at screening
* Clear history of childhood and/or current asthma
* Past history of lung surgery
* Other significant lung disease
* Long term oral steroid treatment
* eGFR < 30 ml/min/1.73 m2 at screening
* NYHA class 3 or 4, where the functional limitation from heart disease is greater than that from COPD, or uncompensated heart failure
* Chronic liver disease (Any elevation of ALT above twice the upper limit of normal at screening. Lower levels of abnormality are permitted after investigator review if felt not to compromise safety)
* Malignancy unless treated and disease free for 5 years
* Conditions causing significant immunosuppression
* Active infection with blood borne viruses (including hepatitis A and B and HIV)
* Other significant medical condition compromising participant safety or fidelity of study.
* Pregnant or breast feeding
* Of childbearing potential and not willing to use highly effective methods of contraception during the course of the study and for 100 days post last dose of mepolizumab.
* Participants who have received an investigational drug within 30 days of first dose, or within 5 drug half-lives of the investigational drug, whichever is longer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in percentage ventilated volume of lung (%VV) | 12 weeks
  The within subject change in percentage ventilated volume of lung (%VV) assessed by XeMRI from baseline to 12 weeks of treatment with mepolizumab
Change in alveolar thickness | 12 weeks
  The within participant change in TP/gas (a measure of alveolar thickness, as an index of pulmonary inflammation) assessed by XeMRI from baseline to 12 weeks of treatment with mepolizumab.

SECONDARY OUTCOMES:
Change in MRI metrics in low and high exacerbation groups | 12 weeks
  Comparison of change in MRI metrics from baseline to 12 weeks in groups with a) low or b) high total 52 week exacerbation (groups defined by median split of total exacerbations over 52 weeks assessed by EXACT-Pro)
Change in MRI indices of ventilation, perfusion and inflammation - 12 weeks | 12 weeks
  Change in MRI indices of ventilation, perfusion and inflammation - CV, RBC/TP, RBC/gas, ADC, LmD, Ve, Ktrans, PBV, PBF, MTT, VQ-intersect, T1, M0 from baseline to 12 weeks

OTHER OUTCOMES:
Change in MRI indices of ventilation, perfusion and inflammation - 52 weeks | 52 weeks
  Change in MRI indices of ventilation, perfusion and inflammation (see text) - %VV, CV, RBC/TP, TP/gas, RBC/gas, ADC, LmD, Ve, Ktrans, PBV, PBF, MTT, VQ-intersect, T1, M0 at 52 weeks compared to baseline and 12 weeks
Correlation of changes to measures of lung function and inflammation (MRI and physiological) | 12 weeks
  Correlation of changes in physiological measures and MRI measures of lung function and inflammation (see text) at 12 weeks
Various correlations of change of ventilation, perfusion and inflammation measures | 12 weeks and 52 weeks
  Change in physiological and MRI determined measures of ventilation, perfusion and inflammation at 12 weeks from baseline will be correlated with;
  1. Baseline peripheral blood eosinophil count
  2. Baseline FeNO
  3. Change of peripheral blood eosinophil count from baseline to 12 weeks
  4. Change in FeNO from baseline to 12 weeks. Similar correlation will be carried out for data obtained at 52 weeks rather than 12 weeks.
Change in MRI metrics in groups with low or high numbers of moderate to severe exacerbations | 12 weeks
  Comparison of change in MRI metrics from baseline to 12 weeks in groups with a) low or b) high total 52 week exacerbation (groups defined by median split of total moderate to severe exacerbations over 52 weeks assessed by EXACT-Pro)
Overall impact of mepolizumab treatment on HRQoL in COPD | 12 and 52 weeks
  Comparison of change of CAT from baseline to 12 and 52 weeks within participants compare to changes in measures of lung function by physiology and MRI.
Overall impact of mepolizumab treatment on HRQoL in COPD | 12 and 52 weeks
  Comparison of changes in physiological and MRI derived parameters at 12 weeks in groups with either high and low improvement of CAT at 52 weeks (determined by median split)
Correlation of PREFUL and DCE MRI measures | 52 weeks (all timepoints)
  PREFUL %VV and PREFUL %PV will be correlated with XeMRI and proton MRI determined measures of lung function at all time points

CONTACTS AND LOCATIONS:
Overall Officials: Rod Lawson, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Clinical Research Facility - NGH, Sheffield, S Yorkshire, United Kingdom